CLINICAL TRIAL: NCT04917991
Title: Comparison Between Olive Oil and Palm Oil-enricHed chOCOlate Spreads (CHOCO) in Healthy Subjects: a Randomized, Double-blind, Cross-over Study
Brief Title: Comparison Between Olive Oil and Palm Oil-enricHed chOCOlate Spreads (CHOCO) in Healthy Subjects
Acronym: CHOCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Silvia Manfrini, Head of the Metabolic Diseases Unit, Campus Bio-Medico University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHOCO study
Record Dates: First submitted 2021-05-28; First posted 2021-06-08 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Healthy Diet
Keywords: Ceramides; insulin resistance; lipids; Visual Analogue Scale; appetite; inflammation
MeSH Terms: conditions — Insulin Resistance; Inflammation

STUDY DESIGN:
Intervention Model Description: Following eligibility assessment, the participants will be be randomized based on a double-blind crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extra Virgin Olive Oil Group (Experimental): Subjects will consume 100 grams of Extra Virgin Olive Oil-enriched chocolate spread for 14 days.
  Interventions: Dietary Supplement: Extra Virgin Olive Oil-enriched chocolate spread
- Palm oil Group (Active Comparator): Subjects will consume 100 grams of palm oil enriched chocolate spread for 14 days.
  Interventions: Dietary Supplement: Palm Oil-enriched chocolate spread

INTERVENTIONS:
Dietary Supplement: Extra Virgin Olive Oil-enriched chocolate spread — the intervention consists in the administration of 100g Extra Virgin Olive Oil-enriched chocolate spread each day for 14 days.
  Arms: Extra Virgin Olive Oil Group
Dietary Supplement: Palm Oil-enriched chocolate spread — the intervention consists in the administration of 100g Palm Oil-enriched chocolate spread each day for 14 days.
  Arms: Palm oil Group

SUMMARY:
This clinical trial aims to investigate if extra virgin olive oil (EVOO) or palm oil enriched chocolate spread snacks consumption lead to differential insulin resistance status in young, healthy subjects. Such effect includes difference in a) plasma ceramides, b) glucose metabolism markers, c) lipid profile, d) inflammatory markers, e) hunger/satiety hormonal markers and visual analogue scale.

DETAILED DESCRIPTION:
Exceeding intake of foods high in palmitic acid, abundant in Palm Oil, has been associated with lipotoxicity, a condition featured by high toxic lipids in the body such as ceramides, which ultimately can lead to insulin resistance and therefore to diabetes and increased cardiometabolic risk through the promotion of atheroma plaque formation.

On the other hand, foods high in oleic acid, rich in extra virgin olive oil EVOO and typical of the Mediterranean diet, has been related to reduced insulin resistance and inflammatory state, with proved protective effects against metabolic diseases such as diabetes, hypercholesterolemia and cardiovascular disease.

Therefore, this clinical trial aims to assess potential metabolic differences in relation to daily consumption of EVOO-enriched chocolate spread in comparison with a Palm oil-enriched chocolate spread.

The investigators, therefore, aimed to evaluate the impact of fourteen days consuming the two different oils added to the same chocolate spread in terms of the composition of plasma ceramides as the primary outcome; and as secondary outcomes, changes in glucose metabolism markers (Glucose, Insulin, HOMA-IR), in LDL, total cholesterol, Triglycerides, HDL levels, in inflammation Markers (CRP, IL-6, TNF-a) and in the appetite-regulating hormones (Leptin, Adiponectin, GLP-1, Ghrelin, PYY and Oxyntomodulin) and in the visual analogue scale (VAS) analysis.

Both chocolate spreads have an identical composition with the exception of fat content (EVOO vs. Palm Oil).

Once eligibility will be assessed through screening and medical anamnesis, twenty healthy subjects will be enrolled and randomized based on a double-blind, controlled, crossover design.

They will undergo a 1-week "run-in diet" phase before the randomization (V1) and the inception of a 14-day interventional diet phase 1. A compliance visit (V2) will be performed on day-7 to ensure that daily compliance is available from each participant (i.e., that the chocolate spread provided is eaten daily). On day 14, the participants will undergo a meal Challenge (V3), consuming the chocolate spread jar (challenge meal) and, serial blood withdrawals will be performed at times 0 ', 30', 60 ', 90', 120 'and 180 ' and, at the same time points, subjects will be required to complete a Visual Analogue Scale (VAS) for monitoring hunger and satiety. Subsequently, the subjects will undergo another week of run-in diet, identical to the previous run-in diet, to be then allocated to another fourteen days of the opposite treatment to the previous one, with the same described methods. Also, in all the visits physical examination with the collection of anthropometric data and body composition analysis will be performed.

Study subjects will be provided structured meals, according to isocaloric diets designed by nutritionists based on subjects' energy requirements. Meals will be prepared by specific canteens and consumed on-site or collected daily in individual meal boxes. Patients will be asked to fill daily food diaries, in order to ensure all of the daily food is ingested (including the chocolate spread), as well as to assess any leftovers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both genders.
* Aged > 18 years.
* Body mass index ranging from 18 to 29.99 kg/m2.
* Subjects able to provide written informed consent.

Exclusion Criteria:

* Diagnosis of diabetes. defined as per the Italian Society of Diabetology guidelines. fasting glucose twice greater than 126 mg / dL and/or random glucose greater than 200 mg / dL.
* Subjects being treated with oral and/or injectable hypoglycemic and/or insulin-sensitizing agents
* Subjects undergoing therapy with synthetic cholesterol-lowering agents (statins and/or fibrates) and/or cholesterol-lowering nutraceuticals (berberine and/or monacolin k)
* Individuals with triglycerides greater than 200 mg/dL
* Subjects with LDL greater than 159 mg/dL
* Moderate or major renal impairment (and GFR <60 mL/min)
* Hypertensive subjects and/or subjects being treated with antihypertensives
* Subjects receiving omega 3 supplements.
* Pregnancy and/or breastfeeding.
* Coronary cardiovascular disease.
* Stroke and heart failure.
* Celiac disease.
* Malabsorption.
* Irritable bowel syndrome.
* Chronic inflammatory bowel disease.
* Present alcoholism or drug abuse or use of medicines whose dose may change during the study or when there is an intention to start a new therapy.
* Individuals with an allergy to hazelnuts or any of the ingredients present in the chocolates under study.
* Neurological or psychiatric pathologies
* Subjects who cannot participate in the study for any reason
* Infectious diseases such as HIV, hepatitis or chronic infections
* Any uncontrolled endocrine pathology such as Cushing's. Acromegaly. etc.
* Any existing cancer and/or lymphoma
* Eating disorders such as anorexia and bulimia
* Previous bariatric surgery or gastrectomy
* Individuals with pacemakers
* Not consuming the chocolate spread for more than three days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 1:1 ratio for the 20 participants enrolled
Enrollment: 20 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Plasma Ceramides | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Fasting Ceramides expressed in nmol

SECONDARY OUTCOMES:
Plasma HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  HOMA-IR calculated as ((fasting insulin (mU/mL) x fasting glucose (mg/dL))/405)
Plasma Insulin | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Fasting Plasma Insulin reported in mU/mL
Plasma Glucose | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Fasting Plasma glucose reported in mg/dL
Plasma Low Density Lipoprotein (LDL) | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Fasting LDL reported in mg/dL
Plasma Triglycerides | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Fasting Triglycerides reported in mg/dL
Plasma Total Cholesterol | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Fasting Total Cholesterol reported in mg/dL
Plasma High Density Lipoprotein (HDL) | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Fasting Plasma HDL
Plasma C-reactive protein (CRP) | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Fasting CRP reported in mg/dL
Plasma Interleukin-6 | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Fasting interleukin-6 reported in pg/mL
Plasma Tumor Necrosis Factor-alpha (TNF-alpha) | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Fasting TNF-alpha reported in pg/mL
Plasma Glucagon Like Peptide-1 (GLP-1) | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  GLP-1 Area Under the Curve calculated below the following time points 0', +30', +60', +90', +120', +180' (minutes following chocolate spread consumption) reported in pg/mL*min.
Plasma Oxyntomodulin | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Oxyntomodulin Area Under the Curve calculated below the following time points 0', +30', +60', +90', +120', +180' (minutes following chocolate spread consumption) reported in pg/mL*min.
Plasma Ghrelin | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Ghrelin Area Under the Curve calculated below the following time points 0', +30', +60', +90', +120', +180' (minutes following chocolate spread consumption) reported in pg/mL*min.
Plasma Peptide YY (PYY) | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  PYY Area Under the Curve calculated below the following time points 0', +30', +60', +90', +120', +180' (minutes following chocolate spread consumption) reported in pg/mL*min.
Plasma Leptin | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Leptin Area Under the Curve calculated below the following time points 0', +30', +60', +90', +120', +180' (minutes following chocolate spread consumption) reported in pg/mL*min.
Plasma Adiponectin | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  Adiponectin Area Under the Curve calculated below the following time points 0', +30', +60', +90', +120', +180' (minutes following chocolate spread consumption) reported in pg/mL*min.
Visual Analogue Scale (VAS) | At the end of the dietary interventional phase (each dietary interventional phase is 14 days)
  VAS Area Under the Curve calculated below the following time points 0', +30', +60', +90', +120', +180' (minutes following chocolate spread consumption) reported in mm*min.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Silvia Manfrini, MD, Principal Investigator — Campus Bio-Medico University of Rome
Locations (1):
- Campus Bio-Medico University of Rome, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No